CLINICAL TRIAL: NCT04430023
Title: Epidemiological and Demographic Data From 150 Patients Diagnosed With Coronavirus Disease 2019 Pneumonia in Intensive Care Unit- a Retrospective, Observational Study in Istanbul, Turkey
Brief Title: Epidemiological and Demographic Data From 150 Patients Diagnosed With Coronavirus Disease 2019 Pneumonia
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, AYŞE SÜRHAN ÇINAR, head of anesthesiology, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: DM3334
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Corona Virus Infection; Pneumonia; Acute Respiratory Failure
Keywords: coronavirus disease 2019; pneumonia
MeSH Terms: conditions — Coronavirus Infections; Pneumonia; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: epidemiological and demographic characteristics — Patients' age, gender, BMI, medical history, symptoms at admission (e.g., cough, fever, myalgia, gastrointestinal symptoms, headache), concomitant diseases (e.g., diabetes mellitus, hypertension, chronic lung disease, cerebrovascular disease, kidney disease, heart disease, cancer, smoking

SUMMARY:
In this study, the investigator examined epidemiological and demographic characteristics, risk factors and 28-day mortality of patients admitted to the intensive care unit with the diagnosis of coronavirus disease 2019 pneumonia.

DETAILED DESCRIPTION:
The patients with intensive care requirements were admitted from emergency department and coronavirus disease 2019 wards to our units. The criteria for intensive care requirement was identified as oxygen saturation<90%, partial oxygen pressure<70 mmHg, respiratory rate> 30/min or PaO2/FiO2(partial oxygen pressure/fraction of inspired oxygen) <300 despite conventional oxygen treatment of 5lt/min. Primary objective was the effect of defined data on 28-day mortality, and secondary objective was the impact of lymphocyte count, lactate dehydrogenase, ferritin, D-dimer and procalcitonin levels, and SOFA(Sequential Organ Failure Assessment) score on prognosis, which are among the risk factors determined by previous studies. All data were evaluated and recorded using the standardized International Severe Acute Respiratory and Emerging Infection Consortium (ISARIC) case report forms, complemented by electronic records of the hospital, nurse observation records, and missing information was completed by telephone interviews with patients' relatives.

ELIGIBILITY:
Inclusion Criteria:

* The study was planned retrospectively, cross-sectionally and observationally with 193 patients hospitalized between 16 March 2020 and 15 May 2020 in five different coronavirus disease 2019 intensive care units in two campuses of our hospital.

Exclusion Criteria:

* Health workers, patients hospitalized less than 24 hours, patients with negative polymerase chain reaction tests, and patients who returned to intensive care unit after discharge were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was planned retrospectively, cross-sectionally and observationally with 193 patients hospitalized between 16 March 2020 and 15 May 2020 in five different coronavirus disease 2019 intensive care units in two campuses of our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
mortality | up to 28 days
  mortality rate
demographic characteristics | up to 28 days
  Patients' age, gender, BMI, medical history

CONTACTS AND LOCATIONS:
Overall Officials: ayse cinar, Principal Investigator — chief of anesthesia department
Locations (1):
- Sisli Etfal Research and Training Hospital, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Result] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Result] Kallet RH. A Comprehensive Review of Prone Position in ARDS. Respir Care. 2015 Nov;60(11):1660-87. doi: 10.4187/respcare.04271. PMID 26493592

DOCUMENTS (2):
  • Study Protocol (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT04430023/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT04430023/SAP_001.pdf